CLINICAL TRIAL: NCT06783504
Title: Effect Of Percutaneous Electrical Nerve Field Stimulation (PENFS) On Symptom Control And Autonomic Nervous System Activity In Patients With Diabetes Mellitus
Brief Title: Effect Of Percutaneous Electrical Nerve Field Stimulation on Symptom Control/Nervous System Activity in Patients w/Diabetes Types 1/2
Acronym: PENFS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Thomas V. Nowak, Professor of Clinical Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18260
Record Dates: First submitted 2024-09-09; First posted 2025-01-20 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Diabetes; Gastroparesis
MeSH Terms: conditions — Diabetes Mellitus; Gastroparesis

STUDY DESIGN:
Intervention Model Description: This is a double blind, randomized, sham controlled study. A total of 30 subjects will be enrolled at Indiana University and another 30 at Ohio State University) with 15 subjects in each arm (PENFS device or Sham (no electrical charge)).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Sham arm will have single blind masking. The participant will not know if they are in the Stimulation arm or the Sham arm; only the coordinator/tech will know the status of the arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ACTIVE (electrical charge) (Active Comparator): The PENFS device is placed behind the patient's left ear and connected to stimulation needles on the auricle. The appliance transmits low-frequency electrical impulses throughout the auricle.
  Interventions: Device: PERCUTANEOUS ELECTRICAL FIELD NERVE STIMULATION
- Sham percutaneous electrical nerve field stimulation (no electrical charge) (Sham Comparator): The PENFS device is placed behind the patient's left ear and connected to stimulation needles on the auricle. The appliance will not transmit any electrical impulses.
  Interventions: Device: Sham percutaneous electrical nerve field stimulation

INTERVENTIONS:
Device: PERCUTANEOUS ELECTRICAL FIELD NERVE STIMULATION — The IB-Stim is a percutaneous electrical nerve field stimulator (PENFS) system intended to be used in patients 11-18 years of age with functional abdominal pain associated with irritable bowel syndrome (IBS). The IB-Stim is intended to be used for 120 hours per week up to 3 consecutive weeks, through application to branches of Cranial Nerves V, VII, IX and X, and the occipital nerves identified by transillumination, as an aid in the reduction of pain when combined with other therapies for IBS.
  Other Names: IB-STIM
  Arms: ACTIVE (electrical charge)
Device: Sham percutaneous electrical nerve field stimulation — SHAM (no electrical charge)
  Other Names: Sham arm
  Arms: Sham percutaneous electrical nerve field stimulation (no electrical charge)

SUMMARY:
The purpose of this study is to find out if we can stimulate the vagus nerve. The vagus nerve is a largely internal nerve that controls many bodily functions, including stomach function. We hope that electrically stimulating the nerve around the external ear will also stimulate the internal vagus nerve. If it does, then we hope that this will help our treatment of patients with nausea and vomiting and disordered stomach function.

DETAILED DESCRIPTION:
Each participant will be randomized to receive Percutaneous Electrical Nerve Field Stimulation (PENFS) treatment with or without stimulation. The study involves 6 study visits. Study procedures include: removing and replacing the PENFS device, questionnaires, ECG, assessment use of galvanic skin response (GSR), pneumatic belt to assess breathing, physical examine, and blood draws.

ELIGIBILITY:
Inclusion Criteria:

* Wiling to have one teaspoon (5 ml) of blood drawn.
* Diagnosed with gastroparesis for twelve months or longer
* Diagnosed with diabetes either Type 1 or Type 2
* Documented delayed gastric emptying (>10% retention of the test meal at four hours) on a standardized scrambled-egg scintigraphy gastric emptying test performed in the last two years.
* Upper GI endoscopy indicating no mechanical obstruction performed in the last five years.
* Symptoms of nausea and vomiting consistent with clinical diagnosis of gastroparesis (as opposed to other causes of nausea and vomiting such as mechanical obstruction, acute viral illness, chemotherapy, psychogenic vomiting.
* Documented Hb A1c within three months of screening or at the time of screening (<=8.0)

Exclusion Criteria:

* Unable to provide consent
* Pregnant females
* Medical records indicate intestinal pseudo-obstruction
* Diagnosed with cardiac arrhythmia
* History of prior gastric surgery
* History of vagotomy
* History of organ transplantation
* History of seizures
* Diagnosed with primary swallowing disorders
* Subjects who are dependent on drugs like Marinol for their condition
* Those diagnosed with psychogenic vomiting and not related to gastroparesis
* Medically unstable subjects
* Those at high surgical risk
* Subjects taking narcotic analgesics daily.
* Those with poorly controlled diabetes mellitus (Hgb A1c>8) within three months of screening or at the time of screening.
* Subjects diagnosed with hemophilia, psoriasis vulgaris are excluded
* Those having a cardiac pacemaker will be excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in Gastroparesis Cardinal Symptom Index Daily Dairy | Five weeks
  ANMS GASTROPARESIS CARDINAL SYMPTOM INDEX - DAILY DIARY this tool uses a list of 7 criteria for rating gastric symptoms. The scale ratings are: None, Mild, Moderate, Severe, and Very Severe.
Change in Patient Assessment of Upper Gastrointestinal Disorder Symptoms | Five weeks
  Scores are calculated by averaging the scores for each item in the subscale, with scores ranging from 0 (none or absent) to 5 (very severe). Optimal outcome would be a score of zero, no episodes/symptoms.

SECONDARY OUTCOMES:
Change in Heart Rate Variability | Five weeks.
  Heart Rate Variability is reported on a 0-100 scale.
Change in Anxiety | Five weeks
  The General Anxiety Disorder (GAD)-7 scale is from 0-21, where 0= no anxiety and 21=severe anxiety
Change in the measure of depression | Five weeks
  Patient Health Questionnaire (PHQ)-8 is a questionnaire that measures self-reported depressive systems. PHQ-8 uses a range from 0-24, where 0=no depressive symptoms and 24=severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas V Nowak, MD, Principal Investigator — IU School of Medicine/IU Health
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
All data and devices will be stored containing only the study subject number and dates of device usage. Sharing this data will not involve any IPD.

REFERENCES:
- [Background] Revicki DA, Speck RM, Lavoie S, Puelles J, Kuo B, Camilleri M, Almansa C, Parkman HP. The American neurogastroenterology and motility society gastroparesis cardinal symptom index-daily diary (ANMS GCSI-DD): Psychometric evaluation in patients with idiopathic or diabetic gastroparesis. Neurogastroenterol Motil. 2019 Apr;31(4):e13553. doi: 10.1111/nmo.13553. Epub 2019 Feb 7. PMID 30734412
- [Background] Kovacic K, Kolacz J, Lewis GF, Porges SW. Impaired Vagal Efficiency Predicts Auricular Neurostimulation Response in Adolescent Functional Abdominal Pain Disorders. Am J Gastroenterol. 2020 Sep;115(9):1534-1538. doi: 10.14309/ajg.0000000000000753. PMID 32732620
- [Background] Berntson GG, Bigger JT Jr, Eckberg DL, Grossman P, Kaufmann PG, Malik M, Nagaraja HN, Porges SW, Saul JP, Stone PH, van der Molen MW. Heart rate variability: origins, methods, and interpretive caveats. Psychophysiology. 1997 Nov;34(6):623-48. doi: 10.1111/j.1469-8986.1997.tb02140.x. PMID 9401419
- [Background] Lewis GF, Furman SA, McCool MF, Porges SW. Statistical strategies to quantify respiratory sinus arrhythmia: are commonly used metrics equivalent? Biol Psychol. 2012 Feb;89(2):349-64. doi: 10.1016/j.biopsycho.2011.11.009. Epub 2011 Dec 3. PMID 22138367
- [Background] Porges SW. Method and apparatus for evaluating rhythmic oscillations in aperiodic physiological response systems. US4510944A, 1985 cited 2020 Aug 4.
- [Background] Asahina M, Poudel A, Hirano S. Sweating on the palm and sole: physiological and clinical relevance. Clin Auton Res. 2015 Jun;25(3):153-9. doi: 10.1007/s10286-015-0282-1. Epub 2015 Apr 17. PMID 25894655
- [Background] 11. Dawson ME, Schell AM, Filion DL. The electrodermal system. In: Handbook of Physiology. 3rd ed. New York: Cambridge University Press; 2007. p. 159-81.
- [Background] Woodbury A, Krishnamurthy V, Gebre M, Napadow V, Bicknese C, Liu M, Lukemire J, Kalangara J, Cui X, Guo Y, Sniecinski R, Crosson B. Feasibility of Auricular Field Stimulation in Fibromyalgia: Evaluation by Functional Magnetic Resonance Imaging, Randomized Trial. Pain Med. 2021 Mar 18;22(3):715-726. doi: 10.1093/pm/pnaa317. PMID 33164085
- [Background] Krasaelap A, Sood MR, Li BUK, Unteutsch R, Yan K, Nugent M, Simpson P, Kovacic K. Efficacy of Auricular Neurostimulation in Adolescents With Irritable Bowel Syndrome in a Randomized, Double-Blind Trial. Clin Gastroenterol Hepatol. 2020 Aug;18(9):1987-1994.e2. doi: 10.1016/j.cgh.2019.10.012. Epub 2019 Oct 14. PMID 31622740
- [Background] Santucci NR, King C, El-Chammas KI, Wongteerasut A, Damrongmanee A, Graham K, Fei L, Sahay R, Jones C, Cunningham NR, Coghill RC. Effect of percutaneous electrical nerve field stimulation on mechanosensitivity, sleep, and psychological comorbidities in adolescents with functional abdominal pain disorders. Neurogastroenterol Motil. 2022 Aug;34(8):e14358. doi: 10.1111/nmo.14358. Epub 2022 Mar 16. PMID 35293081
- [Background] Kovacic K, Hainsworth K, Sood M, Chelimsky G, Unteutsch R, Nugent M, Simpson P, Miranda A. Neurostimulation for abdominal pain-related functional gastrointestinal disorders in adolescents: a randomised, double-blind, sham-controlled trial. Lancet Gastroenterol Hepatol. 2017 Oct;2(10):727-737. doi: 10.1016/S2468-1253(17)30253-4. Epub 2017 Aug 18. PMID 28826627
- [Background] Ward MP, Gupta A, Wo JM, Rajwa B, Furness JB, Powley TL, Nowak TV. An emerging method to noninvasively measure and identify vagal response markers to enable bioelectronic control of gastroparesis symptoms with gastric electrical stimulation. J Neurosci Methods. 2020 Apr 15;336:108631. doi: 10.1016/j.jneumeth.2020.108631. Epub 2020 Feb 20. PMID 32087238
- [Background] Frangos E, Ellrich J, Komisaruk BR. Non-invasive Access to the Vagus Nerve Central Projections via Electrical Stimulation of the External Ear: fMRI Evidence in Humans. Brain Stimul. 2015 May-Jun;8(3):624-36. doi: 10.1016/j.brs.2014.11.018. Epub 2014 Dec 6. PMID 25573069
- [Background] Garcia RG, Lin RL, Lee J, Kim J, Barbieri R, Sclocco R, Wasan AD, Edwards RR, Rosen BR, Hadjikhani N, Napadow V. Modulation of brainstem activity and connectivity by respiratory-gated auricular vagal afferent nerve stimulation in migraine patients. Pain. 2017 Aug;158(8):1461-1472. doi: 10.1097/j.pain.0000000000000930. PMID 28541256
- [Background] Abell T, McCallum R, Hocking M, Koch K, Abrahamsson H, Leblanc I, Lindberg G, Konturek J, Nowak T, Quigley EM, Tougas G, Starkebaum W. Gastric electrical stimulation for medically refractory gastroparesis. Gastroenterology. 2003 Aug;125(2):421-8. doi: 10.1016/s0016-5085(03)00878-3. PMID 12891544